CLINICAL TRIAL: NCT02389244
Title: A Randomized Phase II, Placebo-controlled, Multicenter Study Evaluating Efficacy and Safety of Regorafenib in Patients With Metastatic Bone Sarcomas
Brief Title: A Phase II Study Evaluating Efficacy and Safety of Regorafenib in Patients With Metastatic Bone Sarcomas
Acronym: REGOBONE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UC-0150/1309; 2013-003910-42 (EudraCT Number)
Record Dates: First submitted 2015-02-09; First posted 2015-03-17 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ewing Sarcomas; Chondrosarcomas; Osteosarcomas; Chondroma; CIC-Rearranged Sarcoma
MeSH Terms: conditions — Chondrosarcoma; Osteosarcoma; Chondroma | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regorafenib (Experimental): For adult patients (≥18 years old) : 160 mg/d once daily for the 3 weeks on / 1 week off plus Best Supportive Care (BSC) until progression (according to RECIST 1.1), intolerance or withdrawal of consent .
  For children Age ≥10 years to <18 years old and BSA ≥1.30 m², regorafenib (82 mg/m²) once daily for the 3 weeks on/1 week off (without exceeding 160 mg/day) plus Best Supportive care (BSC) until progression (according to RECIST 1.1), intolerance or withdrawal of consent.
  Interventions: Drug: Regorafenib
- placebo (Placebo Comparator): Placebo plus BCS until progression (according to RECIST V1.1) intolerance or withdrawal of consent. Patients who have received placebo will receive open-label regorafenib after objective tumor progression.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regorafenib — For adults patients and children with BSA ≥1.70 m² : 4 tablets once daily until progression or unacceptable toxicity For children with BSA ≥1.30 and ≤1.69 m² : 3 tablets once daily until progression or unacceptable toxicity
  Other Names: Stivarga
  Arms: Regorafenib
Drug: Placebo — For adults patients and children with BSA ≥1.70 m² : 4 tablets once daily and switch to regorafenib after confirmed progression For children with BSA ≥1.30 and ≤1.69 m² : 3 tablets once daily and switch to regorafenib after confirmed progression
  Other Names: Placebo tablet
  Arms: placebo

SUMMARY:
INDICATION:

Metastatic bone sarcomas: conventional high grade osteosarcoma, Ewing sarcoma of bone, intermediate or high-grade chondrosarcomas and chordomas and either bone or soft tissue metastatic CIC-rearranged sarcomas

DETAILED DESCRIPTION:
METHODOLOGY:

Randomized, placebo-controlled, multicentric, phase II study -This is a double-blind placebo-controlled trial, with 5 cohorts: cohort A: Osteosarcoma, cohort B: Ewing sarcoma, cohort C: Chondrosarcoma, cohort D : chondroma, cohort E: CIC-rearranged sarcoma. Cohort A, B and C will involve a total of 36 patients (24 Regorafenib + 12 placebo), cohort D a total of 24 evaluable patients (16 Regorafenib + 8 placebo) and cohort E will involve a total of 27 evaluable patients (18 Regorafenib + 9 placebo).

159 patients who meet the eligibility criteria will be randomly assigned in a 2:1 ratio to the following treatment groups :

The Arm A:

Regorafenib (160 mg/d) once daily for the 3 weeks on / 1 week off plus Best Supportive Care (BSC) until progression (according to RECIST 1.1), intolerance or withdrawal of consent .

Patients receiving regorafenib who experience disease progression and for whom in the investigator opinion, treatment with regorafenib is providing clinical benefit, may continue the treatment following consultation with the study coordinator and the sponsor.

The Arm B:

Placebo plus BSC until progression (according to RECIST V1.1) intolerance or withdrawal of consent. Patients who have received placebo will receive open-label regorafenib after objective tumor progression.

Patients will be stratified at randomization according to histology .

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed diagnosis of bone sarcoma (osteosarcoma, Ewing sarcoma of bone, chondrosarcoma or chordoma);
2. Patients with confirmed disease progression at study entry;
3. Metastatic disease not amenable to surgical resection or radiation with curative intent;
4. Patients must have measurable disease;
5. Prior treatment :

   at least one, but no more than two prior chemotherapy regimen for metastatic disease for osteosarcoma, chondrosarcoma and Ewing sarcoma; neo-adjuvant /maintenance therapy are not counted towards this requirement. Chordoma not pretreated or with 1 or 2 prior (combination) chemotherapy regimen or with one or two prior molecularly targeted therapy, but no more than 2 prior lines of treatment (whatever the indication) can be included. At least 4 weeks since last chemotherapy (6 weeks in case of nitrosoureas and mitomycin C), immunotherapy or any other pharmacological treatment and/or radiotherapy;
6. Age ≥10 years for osteosarcomas, Ewing sarcomas and chondrosarcomas (for chordomas, patients must be ≥18 years);
7. Body Surface Area ≥1.30 m²;
8. Life expectancy of greater than 3 months;
9. Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky ≥60%) for adults patients;
10. Karnofsky scale ≥ 60% for children aged >12 years old / Lansky scale ≥60% for children aged ≤12 years old;
11. Patients must have adequate bone marrow, renal, and hepatic function, as evidenced by the following within 7 days of study treatment initiation: normal organ function as defined below:

    * Absolute neutrophil count ≥1.5 Giga/L
    * Platelets ≥100 Giga/L
    * Hemoglobin ≥9 g/dL
    * Serum creatinin ≤1.5 x upper limit of normal (ULN)
    * Glomerular filtration rate (GFR) ≥30 ml/min/1.73 m² according to the modified Diet in Renal Disease (MDRD) abbreviated formula
    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x ULN
    * Bilirubin ≤1.5 X ULN
    * Alkaline phosphatase ≤2.5 x ULN (≤5 x ULN in patient with liver involvement of their cancer). If Alkaline phosphatase >2.5 ULN, hepatic isoenzymes 5-nucleotidase or gamma-glutamyl transferase (GGT) tests must be performed; hepatic isoenzymes 5-nucleotidase must be within the normal range and/or GGT <1.5 x ULN;
    * lipase ≤1.5 x ULN;
    * Spot urine must not show 1+ or more protein in urine or the patient will require a repeat urine analysis. If repeat urinalysis shows 1+ protein or more, a 24-hour urine collection will be required and must show total protein excretion <1000 mg/24 hours
12. International Normalized Ratio(INR)/ Partial Thromboplastin Time (PTT) ≤1.5 x ULN;
13. Recovery to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0 Grade 0 or 1 level or recovery to baseline preceding the prior treatment from any previous drug/procedure related toxicity (except alopecia, anemia, and hypothyroidism);
14. Women of childbearing potential and male patients must agree to use adequate contraception for the duration of study participation and up to 3 months following completion of therapy;
15. Women of childbearing potential must have a negative serum β-HCG pregnancy test within 7 days prior randomization and/or urine pregnancy test within 48 hours before the first administration of the study treatment;
16. Signed informed consent form by adult patients and/or patients parents/legal representatives (if age <18 years) and age appropriate assent form by the patients' parents/legal representatives obtained before any study specific procedure is conducted;
17. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures;
18. Patients or parents/legal representatives affiliated to the Social Security System.

Exclusion Criteria:

1. Prior treatment with any VEGFR inhibitor;
2. Soft tissue sarcoma;
3. Other cancer (different histology) within 5 years prior to randomization;
4. Major surgical procedure, open biopsy, significant trauma, within the last 28 days before randomization;
5. Cardiovascular dysfunction:

   * Left ventricular ejection fraction (LVEF) <50%
   * Congestive heart failure (New York Heart Association [NYHA]) ≥2
   * Myocardial infarction <6 months before study
   * Cardiac arrhythmias requiring therapy
   * Uncontrolled hypertension
   * Unstable angina or new-onset angina
6. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within the last 6 months before randomization;
7. Severe hepatic impairment (Child-Pugh C);
8. Ongoing infection > Grade 2 according to NCI-CTCAE v4.0;
9. Known history of human immunodeficiency virus (HIV) infection;
10. Active hepatitis B or C or chronic hepatitis B or C requiring treatment with antiviral therapy;
11. Difficulties with swallowing study tablets;
12. Prior anticancer therapy, including radiotherapy, endocrine therapy, immunotherapy, chemotherapy (CT) within the last 4 weeks (6 weeks for nitrosoureas and mitomycin C), or other investigational agents ; Concomitant antalgic palliative radiotherapy allowed;
13. Concurrent enrolment in another clinical trial in which investigational therapies are administered;
14. Known hypersensitivity to the active substance or to any of the excipients;
15. Pregnant women, women who are likely to become pregnant or are breast-feeding;
16. For adult patients, individual deprived of liberty or placed under the authority of a tutor;
17. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
18. Patients with history of non compliance to medical regimens or unwilling or unable to comply with the protocol;
19. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent;
20. Non-healing wound, non-healing ulcer, or non-healing bone fracture;
21. Patients with evidence or history of any bleeding diathesis, irrespective of severity;
22. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication;
23. Use of biological response modifiers, such as granulocyte colony stimulating factor (G-CSF), within 3 weeks of study entry.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Non-progression rate | 8 weeks for cohorts A, B and E, 12 weeks for cohort C, 6 months for cohort D
  Proportion of patients without disease progression at the defined timepoint after central radiological review (using RECIST 1.1)

SECONDARY OUTCOMES:
Progression Free Survival | expected average duration of 3 months
  from the date of randomization until the date of radiological progression or death whatever the cause (if death occurs before progression)
Objective response rate | 6 months
  complete response (CR) or partial response (PR) according to RECIST 2009, version 1.1, for all cohorts, and CHOI criteria for chordoma
Disease control rate at 6 months | 6 months
  from the date of randomization until the date of death due to any cause
Overall survival | 2 years
  from the date of randomization until the date of death due to any cause
Duration of response | expected average duration of 6 months
  objective response of CR or PR, whichever is noted earlier, to first disease progression or death before progression
Progression-free rate at 3 and 6 months | at 3 and 6 months
  the proportion of patients without progression at 3 and 6 months post randomization
Time to progression | from date of randomization until the date of first observation of progression (up to 6 months)
  from date of randomization until the date of first observation of progression
Growth Modulation Index defined as ratio of time to progressive disease (PD) under regorafenib to time to progression (TTP) under previous treatment | expected average duration of 3 months
  ratio of time to PD under regorafenib to TTP under previous treatment
Toxicity according to NCI-CTCAE V4-0 | expected average duration of 6 months
  according to NCI-CTCAE V4-0 (National Cancer Institut Common Terminology Criteria for Adverse Events)
Pain assessment using Visual analog scale (VAS), DN4 scale (Neuropathic Pain Diagnostic Questionnaire) and NPSI scale (Neuropathic Pain Symptom Inventory) | expected average duration of 6 months
  for chordomas cohort only
PFS | from date of randomization until the date of first observation of progression (up to 6 months)
  Progression Free Survival according to Choi criteria for Chordoma

CONTACTS AND LOCATIONS:
Overall Officials: Florence DUFFAUD, MD PhD, Principal Investigator — La Timone University Hospital
Locations (19):
- France (19):
  - Hopital Jean Monjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - La Timone University Hospital, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin, Paris
  - Institut Curie, Paris
  - Centre Eugene Marquis, Rennes
  - Institut de cancerologie de l'ouest site Rene Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien Neuwirth (ICLN), Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours
  - Institut de cancerologie de lorraine alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
no individual participant data is shared

REFERENCES:
- [Derived] Duffaud F, Italiano A, Bompas E, Rios M, Penel N, Mir O, Piperno-Neumann S, Chevreau C, Delcambre C, Bertucci F, Boudou-Rouquette P, Cancel M, Perrin C, Saada-Bouzid E, Monard L, Schiffler C, Chaigneau L, Hervieu A, Collard O, Bouvier C, Vidal V, Chabaud S, Blay JY; French Sarcoma Group. Efficacy and safety of regorafenib in patients with metastatic or locally advanced chondrosarcoma: Results of a non-comparative, randomised, double-blind, placebo controlled, multicentre phase II study. Eur J Cancer. 2021 Jun;150:108-118. doi: 10.1016/j.ejca.2021.03.039. Epub 2021 Apr 22. PMID 33895682
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- [Derived] Duffaud F, Mir O, Boudou-Rouquette P, Piperno-Neumann S, Penel N, Bompas E, Delcambre C, Kalbacher E, Italiano A, Collard O, Chevreau C, Saada E, Isambert N, Delaye J, Schiffler C, Bouvier C, Vidal V, Chabaud S, Blay JY; French Sarcoma Group. Efficacy and safety of regorafenib in adult patients with metastatic osteosarcoma: a non-comparative, randomised, double-blind, placebo-controlled, phase 2 study. Lancet Oncol. 2019 Jan;20(1):120-133. doi: 10.1016/S1470-2045(18)30742-3. Epub 2018 Nov 23. PMID 30477937